CLINICAL TRIAL: NCT05213897
Title: Clinical Performance Evaluation of SARS-CoV-2 Antigen Assay in Point of Care Settings
Brief Title: Clinical Performance Evaluation of SARS-CoV-2 (COVID-19) Antigen Assay in Point of Care Settings
Status: Completed | Type: Observational
Sponsor: Freedom For All Diagnostics (Industry)
Collaborators: CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: FFA-CV19_1006
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 subjects testing positive for Covid-19: 30 subjects testing positive for Covid-19 using the proprietary SARS-CoV-2 Antigen Assay
  Interventions: Device: SARS-CoV-2 Antigen Assay
- 30 subjects testing negative for Covid-19: 30 subjects testing negative for Covid-19 using the proprietary SARS-CoV-2 Antigen Assay
  Interventions: Device: SARS-CoV-2 Antigen Assay

INTERVENTIONS:
Device: SARS-CoV-2 Antigen Assay — To demonstrate that non-laboratory personnel can accurately perform the SARS-CoV-2 Antigen assay in the intended use environment using nasopharyngeal samples by demonstrating that the assay can achieve a ≥ 80% sensitivity and specificity when it is compared to the results of a high sensitivity EUA SARSCoV-2 RT-PCR assay using nasopharyngeal samples.

SUMMARY:
The purpose of this study is to evaluate the performance of Freedom For All Diagnostics, Inc.'s colloidal gold immune technology SARS-CoV-2 Antigen investigational assay when compared to a high-sensitivity Emergency Use Authorization (EUA) SARS-CoV-2 RT-PCR assay. The study will evaluate the accuracy in the intended use environment of the SARS-CoV-2 antigen assay when testing is conducted in a CLIA-waived setting (e.g., a physician's office or clinic) by non-laboratory personnel serving in a healthcare facility or setting.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate that non-laboratory personnel can accurately perform the SARS-CoV-2 Antigen assay in the intended use environment using nasopharyngeal samples by demonstrating that the assay can achieve a ≥ 80% sensitivity when it is compared to the results of a high sensitivity EUA SARSCoV-2 RT-PCR assay using nasopharyngeal samples. This study is designed as a prospective, blinded study to evaluate the sensitivity and specificity of the SARS-CoV-2 Antigen Assay when non-laboratory personnel conduct testing on Subjects presenting with symptoms of COVID-19.

A minimum of 30 positive and 30 negative samples are required in order to meet EUA submission guidelines. Enrollment will continue until both minimum requirements have been achieved.

ELIGIBILITY:
Inclusion Criteria:

* Subject suspected of having COVID-19 infection and within 7 days of symptom onset. This will include at least one of the following:

  * Fever or chills
  * Cough
  * Shortness of breath or difficulty breathing
  * Fatigue
  * Muscle or body aches
  * Headache
  * New loss of taste or smell
  * Sore throat
  * Congestion or runny nose
* In addition to the above primary symptoms, the Subject might also report nausea, vomiting and/or diarrhea, but these symptoms alone are not sufficient to include the Subject in the study.
* Subject is willing to provide consent/assent.
* Subject is willing to have two (2) nasopharyngeal swabs collected for the study and in the event of inconclusive results, be willing to return to the site to have two (2) more nasopharyngeal swabs

Exclusion Criteria:

To be enrolled in the study, each Subject must not meet:

* Subject unable or unwilling to provide informed consent/assent.
* Subject tested positive for SARS-CoV-2 within the past 3 months.
* Subject has already participated in this study.
* Subject is a vulnerable population and deemed inappropriate for study by site Principal Investigator and/or IRB.

Ages: 2 Years to 94 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients experiencing symptoms and presenting for testing of Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Assay Sensitivity - 80% (versus the EUA SARS-CoV-2 RT-PCR assay) | 48 hours
  SARS-CoV-2 Antigen investigational assay shall have an observed sensitivity of at least 80% when the EUA SARS-CoV-2 RT-PCR assay for nasopharyngeal swabs is used as a reference method.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Geller, MD, Principal Investigator — Centennial Medical Group
Locations (1):
- Centennial Medical, Elkridge, Maryland, United States